CLINICAL TRIAL: NCT02717780
Title: Respiratory Impact of Short Life Agents Used in Balanced Anesthesia on Patients Suffering or Suspected of Obstructive Sleep Apnea (OSA) Syndrome
Brief Title: Short Life Agents in Balanced Anesthesia on Obstructive Sleep Apnea Syndrome
Acronym: DESAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, PD Dr, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CER 192/15
Record Dates: First submitted 2016-03-15; First posted 2016-03-24 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Sleep Apnea Syndromes; Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive | interventions — Fentanyl; Sevoflurane; Remifentanil; Desflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SEVO-FENTA (Active Comparator): Patients scheduled for lower limb surgery will receive a balanced anesthesia with fentanyl and sevoflurane.
  Interventions: Drug: Fentanyl and sevoflurane
- DES-REMI (Experimental): Patients scheduled for lower limb surgery will receive a balanced anesthesia with remifentanil and desflurane.
  Interventions: Drug: Remifentanil and desflurane

INTERVENTIONS:
Drug: Fentanyl and sevoflurane
  Arms: SEVO-FENTA
Drug: Remifentanil and desflurane
  Arms: DES-REMI

SUMMARY:
The investigators aim to assess the respiratory effect of short half-life agents in balanced anesthesia on patients suffering from non-treated or suspected obstructive sleep apnea syndrome (OSA) We will study the impact on OSA of a regimen of remifentanil-desflurane versus a regimen of fentanyl-sevoflurane. Each patient will undergo three respiratory portable polygraphies: the night before the surgery ; the first night following the surgery ; the third night following the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Physical status I - III
* Patient scheduled to undergo lower limb orthopedic surgery
* Patients known for non-treated obstructive sleep apnea or suspected of having an obstructive sleep apnea

Exclusion Criteria:

* Patients known for treated obstructive sleep apnea ;
* Severe respiratory disease (i.e., chronic obstructive pulmonary disease, asthma, pulmonary fibrosis);
* Severe cardiovascular disease
* Chronic use of opiates ≥ 30mg/j morphine eq.
* Chronic use of benzodiazepine
* Inability to consent
* Refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Number of apnea and hypopnea events per hour of sleep (Apnea-Hypopnea index) in supine position | postoperative night 1

SECONDARY OUTCOMES:
Number of obstructive apnea events | postoperative night 1 and night 3
Percentage of time with saturation < 90% | postoperative night 1 and night 3
Mean oxygen saturation | postoperative night 1 and night 3
Total sleep duration | postoperative night 1 and night 3
Percentage of time in supine position | postoperative night 1 and night 3
Number of apnea and hypopnea events per hour of sleep (Apnea-Hypopnea index) in supine position | postoperative night 1 and night 3
Mean amplitude of desaturation (AD%) | postoperative night 1 and night 3
Percentage of time in obstructive apnea | postoperative night 1 and night 3
Percentage of time in central apnea | postoperative night 1 and night 3
Percentage of time in mixt apnea | postoperative night 1 and night 3
Sleep Apnea screening questionnaire (STOP BANG questionnaire) | 24h before surgery
Sleep Apnea screening questionnaire (Berlin questionnaire) | 24h before surgery
Sleep Apnea screening questionnaire (Epworth questionnaire) | 24h before surgery
Sleep Apnea screening questionnaire (NOSAS questionnaire) | 24h before surgery
Pain scores (numeric rating scale, 0-10) | postoperative day 0,1,2 and 3
Postoperative nausea and vomiting (yes/no) | postoperative day 0,1,2 and 3
Pruritus (yes/no) | postoperative day 0,1,2 and 3
Opiate consumption (mg morphine) | postoperative day 0,1,2 and 3
Level of satisfaction (visual analog scale) | postoperative day 3

CONTACTS AND LOCATIONS:
Overall Officials: Eric Albrecht, PD, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- CHUV (Centre Hospitalier Universitaire Vaudois), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Albrecht E, Wegrzyn J, Rossel JB, Bayon V, Heinzer R. Impact of spinal versus general anaesthesia on perioperative obstructive sleep apnoea severity in patients undergoing hip arthroplasty: a post hoc analysis of two randomised controlled trials. Br J Anaesth. 2024 Aug;133(2):416-423. doi: 10.1016/j.bja.2024.04.051. Epub 2024 Jun 10. PMID 38862381